CLINICAL TRIAL: NCT04825977
Title: Risk Stratification of Patients Presenting With Upper Gastrointestinal Bleeding to the Emergency Department Using AIMS65 Score and Red Cell Distribution Width
Acronym: RUGBE
Status: Completed | Type: Observational
Sponsor: Jubilee Mission Medical College and Research Institute (Other)
Responsible Party: Principal Investigator, Dr.Vijay Chanchal A B, Junior Resident, Jubilee Mission Medical College and Research Institute
Other Study IDs: 35/18/IEC/JMMC&RI; CTRI/2019/03/018127 (Registry Identifier: Clinical Trials Registry - India)
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Upper Gastrointestinal Bleeding
Keywords: Emergency Department, Upper GI Bleed, Risk Stratification, Mortality, Red Cell Distribution Width, AIMS65 Score, Receiver Observer Characteristic Curve
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Emergencies | interventions — Erythrocyte Indices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: RISK STRATIFICATION USING AIMS65 SCORE AND RDW — Risk Statification of patients presenting with upper gastrointestinal bleeding to the emergency department using AIMS65 score and Red cell Distribution Width.

SUMMARY:
The rationale of this study in UGIB patients is to assess whether the prediction of mortality and morbidity using AIMS65 score improves when used in combination with RDW in the emergency department setting.

DETAILED DESCRIPTION:
UGIB is a ticking time-bomb and emergency physicians are challenged to accurately assess risk, and aggressively manage patients with gastrointestinal bleeding within the stipulated time in the confines of emergency department. If not managed properly, it is associated with high mortality.

Various clinical prediction scores help in risk stratifying such patients. Among the scores, AIMS65 score is the easy to use score and has good mortality predictive accuracy. RDW, once thought as marker of chronic blood loss has recently been identified as a good prognostic indicator as well as good predictor of mortality in conditions where there is acute blood loss.

Both AIMS65 score and RDW value have been used separately as a predictor of morbidity and mortality in patients with UGIB. But there are not much studies so far evaluating their combined role as marker of predicting mortality as well as high risk among UGIB patients. Hence there is a need for a study to know the predictive value of combination of AIMS6S score and RDW in patients presenting to ED with symptoms of UGIB not been much studies comparing the relationship between RDW and upper GI bleed.

The rationale of this study in UGIB patients is to assess whether the prediction of mortality and morbidity using AIMS65 score improves when used in combination with RDW in the emergency department setting.

ELIGIBILITY:
Inclusion Criteria:

1. All patients presenting to ED with UGIB
2. Age more than 18 years of age

Exclusion Criteria:

1. Patients not consenting to study
2. Patients with known hematological disorders
3. Patients in which endoscopy or blood transfusion is done outside
4. Patients in which RDW value and laboratory parameters required for AIMS65 score are not available.

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adult (>18 years of age) patients presenting with UGIB to the ED of Jubilee Mission Medical College and Research Institute during the 18 months' time period were included in the study. The diagnosis of UGIB was based on patients' presentations, including coffee ground vomitus, hematemesis, melena, and blood in nasogastric aspirate. These patients were considered eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 348 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
predictive accuracy of addition of RDW to AIMS65 SCORE in determining the 30-day mortality of patients presenting to the ED with symptoms of UGIB | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Siju V Abraham, MD, Study Chair — Jubilee Mission Medical College; Rajeev P C, MD, Study Director — Jubilee Mission Medical College
Locations (1):
- Jubilee Mission Medical College and Research Institute, Thrissur, Kerala, India